CLINICAL TRIAL: NCT02868502
Title: The Effect of Trabeculectomy, Glaucoma Drainage Device, Cyclophotocoagulation, and Ocular Hypotensive Eye-drops on Intraocular Pressure Fluctuation With Postural Change in Eyes With Open-angle Glaucoma
Brief Title: Different Glaucoma Treatments Effect on Intraocular Pressure Fluctuation With Postural Change in Eyes With Open-angle Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Avner Belkin, MD, Meir Medical Center
Other Study IDs: MMC-0026-16
Record Dates: First submitted 2016-07-27; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Open Angle Glaucoma
Keywords: Glaucoma; Open Angle Glaucoma; Intra Ocular Pressure; Ocular Hypotensive Drops; Trabeculectomy; Cyclophotocoagulation; Glaucoma Drainage Device
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Trabeculectomy: Subjects with OAG s/p Trabeculectomy. IOP measurement in different positions.
  Interventions: Device: Goldmann tonometer; Device: Pneumatonometer; Device: Tonopen XL; Device: ICare rebound tonometer
- Ahmed Glaucoma Valve implantation: Subjects with OAG s/p Ahmed valve implantation. IOP measurement in different positions.
  Interventions: Device: Goldmann tonometer; Device: Pneumatonometer; Device: Tonopen XL; Device: ICare rebound tonometer
- Cyclophotocoagulation: Subjects with OAG s/p Cyclophotocoagulation. IOP measurement in different positions.
  Interventions: Device: Goldmann tonometer; Device: Pneumatonometer; Device: Tonopen XL; Device: ICare rebound tonometer
- Ocular hypotensive eye drops: Subjects with OAG treated with ocular hypotensive eye drops and no ocular surgical hypotensive treatments.
  IOP measurement in different positions.
  Interventions: Device: Goldmann tonometer; Device: Pneumatonometer; Device: Tonopen XL; Device: ICare rebound tonometer
- Ocular Hypertension: Subjects with no evidence of glaucomatous damage, but with IOP measurements above 21 mmHg..
  IOP measurement in different positions.
  Interventions: Device: Goldmann tonometer; Device: Pneumatonometer; Device: Tonopen XL; Device: ICare rebound tonometer
- Control: Subjects with healthy eyes, apart for refraction errors, post cataract surgery, strabismus or amblyopia.
  IOP measurement in different positions.
  Interventions: Device: Goldmann tonometer; Device: Pneumatonometer; Device: Tonopen XL; Device: ICare rebound tonometer

INTERVENTIONS:
Device: Goldmann tonometer — IOP measurement in the sitting position and lateral decubitus
Device: Pneumatonometer — IOP measurement in the sitting position and lateral decubitus
Device: Tonopen XL — IOP measurement in the sitting position and lateral decubitus
Device: ICare rebound tonometer — IOP measurement in the sitting position and lateral decubitus

SUMMARY:
The purpose of this study is to investigate the effect of trabeculectomy, glaucoma drainage devices, cyclophotocoagulation and ocular hypotensive eye-drops on IOP elevation with postural change from the sitting to supine positions in eyes with open-angle glaucoma.

Patients will be assigned to the different study groups according to their past ocular history. Interventions are similar to all study group and no medical therapy alteration will be made.

DETAILED DESCRIPTION:
Visual impairment and blindness due to chronic progressive optic neuropathy developing from glaucoma are major health problems worldwide.

Glaucoma is a progressive, potentially blinding disease, in which the only modifiable risk factor in intraocular pressure. In a significant proportion of patients, the disease progresses despite apparent IOP control(1-3).

One factor which may explain some of this discrepancy is a fluctuation of the IOP during the day, which may be missed in a single visit to the ophthalmologist(4). Although this fluctuation depends to some degree on daily biologic rhythms and the specific type of glaucoma, a constant significant factor responsible for this effect is the IOP-dependent changes of body posture, from sitting or standing to lying down(5). Older studies have shown IOP postural changes in the range of 4-6 mmHg(6-8). Seeing how a typical patient may spend as much as a third of his life in the supine position, knowledge of IOP in this position, and its control, are of great importance in decreasing the chance for irreversible optic nerve damage.

Several studies of Liu JH(9-11) have investigated the effect of hypotensive drops on nocturnal IOP. While prostaglandin analogues (PGA) and carbonic anhydrase inhibitors (CAI) seemed to have a significant nocturnal IOP lowering effect, the effect seen with beta blockers and alpha agonists was minimal. Mansouri et al.(12) recently showed that PGA seem to ﬂatten the IOP-related increase when moving from the sitting to the supine position at nocturnal period, without effecting other circadian IOP-related patterns.

Hirooka Kazuyuki investigated the effect of trabeculectomy on the IOP fluctuations caused by postural changes(13-14). He showed that successful trabeculectomy, which didn't require needling, have significantly decreased the posture-induced IOP changes to less than 3 mmHg.

To the best of our knowledge there is no data regarding the effect of glaucoma drainage devices and cyclophotocoagulation on supine IOP.

The purpose of this study is to investigate the effect of different IOP lowering methods, including trabeculectomy, glaucoma drainage devices, cyclophotocoagulation and ocular hypotensive eye-drops on IOP with postural change from the sitting to supine positions in eyes with open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* OAG patients
* Ocular Hypertension (OHT) patients
* Healthy subjects, without any ocular pathology (except for refraction errors, past cataract surgery, strabismus or amblyopia).

Exclusion Criteria:

* Other intraocular surgeries within the past 3 months
* Illness effecting episcleral venous pressure, such as superior vena cava syndrome, thyroid eye disease, orbital masses
* Patients who are unable to maintain supine position for 15 minutes
* Corneal abnormalities: epithelial pathologies, corneal infection, corneal erosions, corneal scars, keratoconus, S/P corneal transplantation (lamellar/full thickness)
* Hypersensitivity to oxybuprocaine hydrochloride

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects with open angle glaucoma with past ocular history of surgical treatment (trabeculectomy, implantation of an Ahmed glaucoma drainage device or cyclophotocoagulation) or are using ocular hypotensive eye drops and subjects with ocular hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Measurements of Intra Ocular Pressure Fluctuation with Postural Change in Eyes with Open-angle Glaucoma and Ocular Hypertension, compared to healthy subjects | Change from baseline 5 minutes following position change
  Interventions are similar for all study groups: The subject will be instructed to stay in a sitting position for 5 minutes. A topical anesthetic eye drop (oxybuprocaine hydrochloride 0.4%) will then be installed in the study eye (necessary procedure made in all IOP examinations as a regular procedure) and the IOP will be measured, in the following order by 4 tonometers: Goldmann tonometer, Pneumatonometer, Tonopen XL, ICare rebound tonometer. The subject will then lie supine for 5 minutes, afterwards will turn to the lateral decubitus position and IOP will be measured again using the same tonometers in the same manner.
  The difference between IOP in the sitting and lying body positions will be assessed and compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Avner Belkin, M.D, Principal Investigator — Meir Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schulzer M, Mikelberg FS, Drance SM. Some observations on the relation between intraocular pressure reduction and the progression of glaucomatous visual loss. Br J Ophthalmol. 1987 Jul;71(7):486-8. doi: 10.1136/bjo.71.7.486. PMID 3651360
- [Background] Flammer J, Robert Y, Gloor B. Influence of pindolol and timolol treatment on the visual fields of glaucoma patients. J Ocul Pharmacol. 1986 Fall;2(4):305-11. doi: 10.1089/jop.1986.2.305. PMID 3503114
- [Background] Kidd MN, O'Connor M. Progression of field loss after trabeculectomy: a five-year follow-up. Br J Ophthalmol. 1985 Nov;69(11):827-31. doi: 10.1136/bjo.69.11.827. PMID 4063249
- [Background] Barkana Y, Anis S, Liebmann J, Tello C, Ritch R. Clinical utility of intraocular pressure monitoring outside of normal office hours in patients with glaucoma. Arch Ophthalmol. 2006 Jun;124(6):793-7. doi: 10.1001/archopht.124.6.793. PMID 16769832
- [Background] Barkana Y, Gutfreund S. Measurement of the difference in intraocular pressure between the sitting and lying body positions in healthy subjects: direct comparison of the Icare Pro with the Goldmann applanation tonometer, Pneumatonometer and Tonopen XL. Clin Exp Ophthalmol. 2014 Sep-Oct;42(7):608-14. doi: 10.1111/ceo.12272. Epub 2014 Jan 13. PMID 24299102
- [Background] Weber AK, Price J. Pressure differential of intraocular pressure measured between supine and sitting position. Ann Ophthalmol. 1981 Mar;13(3):323-6. PMID 7258940
- [Background] Buchanan RA, Williams TD. Intraocular pressure, ocular pulse pressure, and body position. Am J Optom Physiol Opt. 1985 Jan;62(1):59-62. doi: 10.1097/00006324-198501000-00008. PMID 3976837
- [Background] Yamabayashi S, Aguilar RN, Hosoda M, Tsukahara S. Postural change of intraocular and blood pressures in ocular hypertension and low tension glaucoma. Br J Ophthalmol. 1991 Nov;75(11):652-5. doi: 10.1136/bjo.75.11.652. PMID 1751457
- [Background] Liu JH, Kripke DF, Weinreb RN. Comparison of the nocturnal effects of once-daily timolol and latanoprost on intraocular pressure. Am J Ophthalmol. 2004 Sep;138(3):389-95. doi: 10.1016/j.ajo.2004.04.022. PMID 15364220
- [Background] Liu JH, Medeiros FA, Slight JR, Weinreb RN. Diurnal and nocturnal effects of brimonidine monotherapy on intraocular pressure. Ophthalmology. 2010 Nov;117(11):2075-9. doi: 10.1016/j.ophtha.2010.03.026. Epub 2010 Jul 21. PMID 20663566
- [Background] Tung JD, Tafreshi A, Weinreb RN, Slight JR, Medeiros FA, Liu JH. Twenty-four-hour effects of bimatoprost 0.01% monotherapy on intraocular pressure and ocular perfusion pressure. BMJ Open. 2012 Aug 23;2(4):e001106. doi: 10.1136/bmjopen-2012-001106. Print 2012. PMID 22918671
- [Background] Mansouri K, Medeiros FA, Weinreb RN. Effect of glaucoma medications on 24-hour intraocular pressure-related patterns using a contact lens sensor. Clin Exp Ophthalmol. 2015 Dec;43(9):787-95. doi: 10.1111/ceo.12567. Epub 2015 Aug 16. PMID 26152693
- [Background] Hirooka K, Takenaka H, Baba T, Takagishi M, Mizote M, Shiraga F. Effect of trabeculectomy on intraocular pressure fluctuation with postural change in eyes with open-angle glaucoma. J Glaucoma. 2009 Dec;18(9):689-91. doi: 10.1097/IJG.0b013e31819c49f4. PMID 20010249
- [Background] Hirooka K, Tenkumo K, Nitta E, Sato S. Correlation between Intraocular Pressure Fluctuation with Postural Change and Postoperative Intraocular Pressure in Relation to the Time Course after Trabeculectomy. J Ophthalmol. 2014;2014:801967. doi: 10.1155/2014/801967. Epub 2014 Jul 17. PMID 25136454